CLINICAL TRIAL: NCT02528318
Title: A Multicenter, Randomized, Open-label, Controlled Trial To Assess The Safety And Tolerability Of Lucinactant For Inhalation In Preterm Neonates 26 to 28 Weeks PMA
Brief Title: Trial To Assess The Safety And Tolerability Of Lucinactant For Inhalation In Preterm Neonates 26 to 28 Weeks PMA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to terminate after 3 dosing groups
Sponsor: Windtree Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 03-CL-1401
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — lucinactant; Inhalation; Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 50 mg/kg (Experimental): Lucinactant for inhalation 50 mg total phospholipids (TPL)/kg with nCPAP
  1 repeat dose allowed if repeat dosing criteria are met.
  Interventions: Combination Product: Lucinactant for inhalation
- 75 mg/kg (Experimental): Lucinactant for inhalation 75 mg TPL/kg with nCPAP
  1 repeat dose allowed if repeat dosing criteria are met.
  Interventions: Combination Product: Lucinactant for inhalation
- 100 mg/kg (Experimental): Lucinactant for inhalation 100 mg TPL/kg with nCPAP
  1 repeat dose allowed if repeat dosing criteria are met.
  Interventions: Combination Product: Lucinactant for inhalation
- 150 mg/kg (Experimental): Lucinactant for inhalation 150 mg TPL/kg with nCPAP
  1 repeat dose will be allowed if repeat dosing criteria are met.
  Interventions: Combination Product: Lucinactant for inhalation
- nCPAP alone (Active Comparator): nCPAP therapy alone
  Interventions: Device: nCPAP alone

INTERVENTIONS:
Combination Product: Lucinactant for inhalation — Lucinactant for inhalation refers to the active investigational agent, lucinactant, in combination with the investigational delivery device (drug-device combination product)
  Other Names: AEROSURF®
  Arms: 100 mg/kg; 150 mg/kg; 50 mg/kg; 75 mg/kg
Device: nCPAP alone — nCPAP therapy
  Other Names: nasal continuous positive airway pressure
  Arms: nCPAP alone

SUMMARY:
This study is to evaluate the safety and tolerability of lucinactant for inhalation, administered as an aerosol in up to four escalating doses to preterm neonates 26 to 28 weeks gestational age who are receiving nCPAP for RDS compared to neonates receiving nCPAP alone.

DETAILED DESCRIPTION:
This study was a multicenter, randomized, controlled, open-label, dose-escalation study, conducted to evaluate the safety and tolerability of lucinactant for inhalation in conjunction with nasal continuous positive airway pressure (nCPAP) in comparison with nCPAP alone. The study was to evaluate the safety and tolerability of lucinactant for inhalation, administered as an aerosol in 4 escalating doses.

For this study, lucinactant for inhalation refers to the active investigational agent, lyophilized lucinactant, in combination with the prototype investigational delivery device. Reconstituted lyophilized lucinactant was aerosolized by the investigational device and introduced into the nCPAP circuit. Those randomized to the control arm continued to receive nCPAP alone. Dose assignments were unblinded, as the primary objective of this study was safety and tolerability.

Preterm neonates with respiratory distress syndrome (RDS) between 26 and 28 completed weeks PMA who were within the first 20 hours after birth and who had successful implementation of controlled nCPAP within 90 minutes of birth were considered to be potential subjects. Before study enrollment, legal guardians were provided a written informed consent form (ICF) for each potential subject.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent from a legally authorized representative.
2. Gestational age 26 to 28 completed weeks post menstrual age (PMA).
3. Successful implementation of controlled nCPAP within 90 minutes after birth.
4. Spontaneous breathing.
5. Chest radiograph consistent with RDS.
6. Within the first 20 hours after birth, have an nCPAP of 5 to 6 cm H2O to maintain oxygen saturation measured by pulse oximetry (SpO2) of 88% to 95% with a fraction of inspired oxygen (FiO2) of 0.25 to 0.50 that is clinically indicated for at least 30 minutes. Transient (<10 minutes) FiO2 excursions below 0.25 or above 0.50 did not reset the 30 minute requirement.

Exclusion Criteria:

1. Heart rate that cannot be stabilized above 100 beats/minute within 5 minutes of birth.
2. Recurrent episodes of apnea occurring after the initial newborn resuscitation period (ie, 10 minutes after birth) requiring intermittent positive pressure breaths using inflating pressures above the set CPAP pressure administered manually or mechanically through any patient interface.
3. A 5 minute Apgar score < 5.
4. Major congenital malformation(s) and cranial/facial abnormalities that preclude nCPAP, diagnosed antenatally or immediately after birth.
5. Other diseases or conditions potentially interfering with cardiopulmonary function (eg, hydrops fetalis or congenital infection such as TORCH).
6. Known or suspected chromosomal abnormality or syndrome.
7. Premature rupture of membranes (PROM) > 2 weeks.
8. Evidence of hemodynamic instability requiring vasopressors or steroids for hemodynamic support and/or presumed clinical sepsis.
9. Need for endotracheal intubation and mechanical ventilation.
10. Has been administered: another investigational agent or investigational medical device, any other surfactant agent, steroid treatment after birth.

Ages: 26 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Simonson, MD, Study Director — Windtree Therapeutics
Locations (20):
- United States (10):
  - Loma Linda University Medical Center, Loma Linda, California
  - Sharp Mary Birch Hospital for Women and Newborns, San Diego, California
  - Christiana Care Health System, Newark, Delaware
  - University of Miami, Miami, Florida
  - University of Louisville, Louisville, Kentucky
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Columbia University College of Physicians and Surgeons, New York Presbyterian Hospital - Morgan Stanley Children's Hospital, New York, New York
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Women and Infants Hospital, Providence, Rhode Island
- Canada (4):
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Alexandria Hospital, Edmonton, Alberta
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
- Chile (2):
  - Hospital Dr Sotero Del Rio, Santiago
  - Hospital San Juan de Dios, Santiago
- Poland (4):
  - Ginekologiczno-Polozniczy Szpital Klinicznym UM im. Karola Marcinkowskiego w Poznan i u Katedra Neonatologii, Poznan, Greater Poland Voivodeship
  - S.U. nr2im. Dr. Jana Biziela Oddzial Kliniczny N. W. Z. Intensywna Terapia Noworodka wraz z Wgjazdowy m Zespolem N, Bydgoszcz, Kujawsko-pomorksie
  - Szpital Kliniczny im. Ks, Anny Mazowieckiej Klinika Neonatologii, Warsaw, Masovian Voivodeship
  - Instytut Centrum Zdrowja Matki Polki Klinika Neonatologii, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 50 mg/kg: Lucinactant for inhalation 50 mg total phospholipids (TPL)/kg with nCPAP
  1 repeat dose allowed if repeat dosing criteria are met.
  Lucinactant for inhalation: Lucinactant for inhalation refers to the active investigational agent, lucinactant, in combination with the investigational delivery device (drug-device combination product)
- 75 mg/kg: Lucinactant for inhalation 75 mg TPL/kg with nCPAP
  1 repeat dose allowed if repeat dosing criteria are met.
  Lucinactant for inhalation: Lucinactant for inhalation refers to the active investigational agent, lucinactant, in combination with the investigational delivery device (drug-device combination product)
- 100 mg/kg: Lucinactant for inhalation 100 mg TPL/kg with nCPAP
  1 repeat dose allowed if repeat dosing criteria are met.
  Lucinactant for inhalation: Lucinactant for inhalation refers to the active investigational agent, lucinactant, in combination with the investigational delivery device (drug-device combination product)
- 150 mg/kg: Lucinactant for inhalation 150 mg TPL/kg with nCPAP
  1 repeat dose will be allowed if repeat dosing criteria are met.
  Lucinactant for inhalation: Lucinactant for inhalation refers to the active investigational agent, lucinactant, in combination with the investigational delivery device (drug-device combination product)
Period: Overall Study
Arm/Group | 50 mg/kg | 75 mg/kg | 100 mg/kg | 150 mg/kg | nCPAP Alone
Started | 8 | 8 | 8 | 0 (Study was terminated prior to initiation of this intervention) | 24
Completed | 8 | 8 | 8 | 0 | 24
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This dose-escalation study was terminated after completion of the 100 mg/kg group for administrative purposes. No participants were enrolled in the 150 mg/kg group or received 150 mg/kg.
Groups:
- 50 mg/kg: Lucinactant for inhalation 50 mg TPL/kg with nCPAP
  1 repeat dose allowed if repeat dosing criteria are met.
  Lucinactant for inhalation: Lucinactant for inhalation refers to the active investigational agent, lucinactant, in combination with the investigational delivery device (drug-device combination product)
- Total: Total of all reporting groups
Arm/Group | 50 mg/kg | 75 mg/kg | 100 mg/kg | 150 mg/kg | nCPAP Alone | Total
Number analyzed (Participants) | 8 | 8 | 8 | 0 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 8 | 8 | 0 | 24 | 48
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Customized [Mean (Standard Deviation); unit: weeks] — Gestational age, based on obstetrician's best estimate
  weeks
    Gestational Age | 27.6 (0.61) | 27.2 (1.06) | 27.2 (0.84) |  | 27.5 (0.76) | 27.4 (0.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 5 |  | 8 | 21
  Male | 5 | 3 | 3 |  | 16 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 2 |  | 7 | 13
  Not Hispanic or Latino | 5 | 7 | 6 |  | 17 | 35
  Unknown or Not Reported | 0 | 0 | 0 |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  | 0 | 0
  Asian | 2 | 0 | 1 |  | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  | 0 | 0
  Black or African American | 1 | 1 | 2 |  | 1 | 5
  White | 3 | 5 | 4 |  | 20 | 32
  More than one race | 0 | 0 | 0 |  | 0 | 0
  Unknown or Not Reported | 2 | 2 | 1 |  | 2 | 7
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 3 | 4 |  | 8 | 16
  United States | 7 | 3 | 4 |  | 12 | 26
  Poland | 0 | 2 | 0 |  | 3 | 5
  Chile | 0 | 0 | 0 |  | 1 | 1
Birth Weight [Mean (Standard Deviation); unit: g] | 1052 (174.7) | 855 (84.6) | 839 (224.9) |  | 1005 (238.8) | 960 (209.4)
Apgar Score at One Minute [Mean (Full Range); unit: Scores on a scale] — The Apgar Score measures a baby's health by assessing five characteristics (Appearance, Pulse, Grimace, Activity, and Respiration) . Each of the five characteristics are scored from 0 to 2, and the five scores are summed for the Apgar Score. Thus, the Apgar Score ranges from 0 (worst) to 10 (best), and scores over 7 indicate a baby in good health. Apgar Scores are performed at 1 minute and 5 minutes after birth.
  Scores on a scale | 5.4 [2 to 9] | 5.5 [2 to 8] | 6.4 [3 to 8] |  | 5.8 [1 to 9] | 5.8 [1 to 9]
Apgar Score at Five Minutes [Mean (Full Range); unit: Scores on a scale] — The Apgar Score measures a baby's health by assessing five characteristics (Appearance, Pulse, Grimace, Activity, and Respiration) . Each of the five characteristics are scored from 0 to 2, and the five scores are summed for the Apgar Score. Thus, the Apgar Score ranges from 0 (worst) to 10 (best), and scores over 7 indicate a baby in good health. Apgar Scores are performed at 1 minute and 5 minutes after birth.
  Scores on a scale | 7.8 [7 to 9] | 6.4 [1 to 9] | 8.1 [6 to 9] |  | 7.9 [5 to 9] | 7.7 [1 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Peri-Dosing Adverse Events - Initial Dose
Description: Number of Participants with adverse events that were experienced during the initial study treatment
Time Frame: Randomization to 24 Hours Post Randomization
Population: Safety Population. Peri-dosing events are events that occur during study treatment. Since this was an open-label study, no peri-dosing events were recorded for nCPAP alone. Any adverse events that occurred during the corresponding time for nCPAP alone were recorded as adverse events but not peri-dosing events.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg/kg | 75 mg/kg | 100 mg/kg | 150 mg/kg | nCPAP Alone
Number analyzed (Participants) | 8 | 8 | 8 | 0 | 0
Participants
  Bradycardia | 0 | 2 | 1 |  |
  Desaturation | 1 | 2 | 3 |  |
  Gagging/regurgitation | 0 | 0 | 0 |  |
  Apnea | 1 | 1 | 1 |  |
  Pallor | 0 | 0 | 0 |  |

2. Primary Outcome: Number of Participants With Air Leak
Description: Number of participants with air leak (includes pneumothorax, pulmonary interstitial emphysema (PIE), pneumomediastinum, pneumopericardium, subcutaneous emphysema)
Time Frame: 7 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg/kg | 75 mg/kg | 100 mg/kg | 150 mg/kg | nCPAP Alone
Number analyzed (Participants) | 8 | 8 | 8 | 0 | 24
Participants | 3 | 0 | 2 |  | 4

3. Secondary Outcome: Number of Participants With Worsening of Respiratory Status Criteria
Description: Number of participants with worsening in one of 12 respiratory status criteria through 72 hours post randomization (need for additional surfactant therapy, desaturation < 80%, heart rate < 100 bpm, sustained fraction of inspired oxygen (FiO2) > 0.50, arterial carbon dioxide (PCO2) > 65 mmHg, sustained apnea, persistent arterial pH < 7.2, intubation for any reason, nCPAP > 7 cmH2O, initiation of intermittent positive pressure ventilation, death, principal investigator determination of worsening status)
Time Frame: Randomization to 72 Hours Post Randomization
Population: Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg/kg | 75 mg/kg | 100 mg/kg | 150 mg/kg | nCPAP Alone
Number analyzed (Participants) | 8 | 8 | 8 | 0 | 24
Participants | 6 | 7 | 6 |  | 18

4. Secondary Outcome: Bronchopulmonary Dysplasia
Description: Number of participants with bronchopulmonary dysplasia (BPD) and number of participants alive and without BPD at 36 weeks post-menstrual age (PMA)
Time Frame: Randomization to 36 weeks PMA
Population: Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg/kg | 75 mg/kg | 100 mg/kg | 150 mg/kg | nCPAP Alone
Number analyzed (Participants) | 8 | 8 | 8 | 0 | 24
Participants
  BPD | 0 | 0 | 0 |  | 6
  Alive and Without BPD | 7 | 7 | 8 |  | 18

5. Secondary Outcome: Number of Participants With Nasal Continuous Positive Airway Pressure (nCPAP) Failure
Description: Participants who required intubation for mechanical ventilation or surfactant administration were defined as having failed nCPAP
Time Frame: Randomization to 72 Hours Post Randomization
Population: Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg/kg | 75 mg/kg | 100 mg/kg | 150 mg/kg | nCPAP Alone
Number analyzed (Participants) | 8 | 8 | 8 | 0 | 24
Participants | 5 | 7 | 5 |  | 16

6. Secondary Outcome: Death
Description: Number of participants who died during the study
Time Frame: Randomization to 36 weeks PMA
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg/kg | 75 mg/kg | 100 mg/kg | 150 mg/kg | nCPAP Alone
Number analyzed (Participants) | 8 | 8 | 8 | 0 | 24
Participants | 1 | 1 | 0 | 0 | 0

7. Secondary Outcome: FiO2
Description: Observed and change from baseline measurements for fraction of inspired oxygen (FiO2). Values represent the amount (fraction) of oxygen in the air the participant inspires; the values themselves do not have units. The normal amount of oxygen in air ("room air") is 21%, or 0.21.
Time Frame: Randomization to 72 hours post randomization
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Fraction of oxygen in inspired air
Arm/Group | 50 mg/kg | 75 mg/kg | 100 mg/kg | 150 mg/kg | nCPAP Alone
Number analyzed (Participants) | 8 | 8 | 8 | 0 | 24
Fraction of oxygen in inspired air
  Baseline (Randomization): number analyzed (Participants) | 8 | 7 | 8 | 0 | 24
  Baseline (Randomization) | 0.31 (0.058) | 0.33 (0.071) | 0.37 (0.072) |  | 0.32 (0.061)
  60 Minutes Post Randomization - Observed: number analyzed (Participants) | 7 | 7 | 7 | 0 | 23
  60 Minutes Post Randomization - Observed | 0.31 (0.064) | 0.35 (0.063) | 0.37 (0.090) |  | 0.34 (0.159)
  60 Minutes Post Randomizati - Change from Baseline: number analyzed (Participants) | 7 | 7 | 7 | 0 | 23
  60 Minutes Post Randomizati - Change from Baseline | 0.01 (0.010) | 0.02 (0.024) | 0.01 (0.044) |  | 0.01 (0.162)
  3 Hours Post Randomization - Observed: number analyzed (Participants) | 8 | 8 | 8 | 0 | 23
  3 Hours Post Randomization - Observed | 0.37 (0.191) | 0.37 (0.120) | 0.37 (0.107) |  | 0.29 (0.082)
  3 Hours Post Randomizaiton - Change from Baseline: number analyzed (Participants) | 8 | 7 | 8 | 0 | 23
  3 Hours Post Randomizaiton - Change from Baseline | 0.06 (0.154) | 0.00 (0.066) | 0.00 (0.047) |  | -0.03 (0.082)
  12 Hours Post Randomization - Observed: number analyzed (Participants) | 8 | 8 | 8 | 0 | 23
  12 Hours Post Randomization - Observed | 0.30 (0.114) | 0.30 (0.117) | 0.30 (0.068) |  | 0.33 (0.181)
  12 Hours Post Randomization - Change from Baseline: number analyzed (Participants) | 8 | 7 | 8 | 0 | 23
  12 Hours Post Randomization - Change from Baseline | -0.02 (0.137) | -0.07 (0.074) | -0.08 (0.090) |  | 0.00 (0.172)
  24 Hours Post Randomized - Observed: number analyzed (Participants) | 8 | 8 | 7 | 0 | 24
  24 Hours Post Randomized - Observed | 0.28 (0.093) | 0.25 (0.044) | 0.28 (0.077) |  | 0.29 (0.143)
  24 Hours Post Randomized - Change from Baseline: number analyzed (Participants) | 8 | 7 | 7 | 0 | 24
  24 Hours Post Randomized - Change from Baseline | -0.03 (0.072) | -0.09 (0.046) | -0.08 (0.105) |  | -0.04 (0.140)
  48 Hours Post Randomized - Observed | 0.28 (0.058) | 0.24 (0.038) | 0.29 (0.071) |  | 0.31 (0.188)
  48 Hours Post Randomized - Change from Baseline: number analyzed (Participants) | 8 | 7 | 8 | 0 | 24
  48 Hours Post Randomized - Change from Baseline | -0.03 (0.083) | -0.09 (0.075) | -0.09 (0.091) |  | -0.02 (0.191)
  72 Hours Post Randomized - Observed: number analyzed (Participants) | 7 | 8 | 8 | 0 | 23
  72 Hours Post Randomized - Observed | 0.30 (0.105) | 0.23 (0.023) | 0.25 (0.050) |  | 0.27 (0.119)
  72 Hours Post Randomized - Change from Baseline: number analyzed (Participants) | 7 | 7 | 8 | 0 | 23
  72 Hours Post Randomized - Change from Baseline | -0.02 (0.133) | -0.10 (0.071) | -0.12 (0.066) |  | -0.05 (0.133)

8. Secondary Outcome: Number of Participants With Complications of Prematurity
Description: Number of participants with pre-specified common complications of prematurity.
Time Frame: Randomization to 36 weeks PMA
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg/kg | 75 mg/kg | 100 mg/kg | 150 mg/kg | nCPAP Alone
Number analyzed (Participants) | 8 | 8 | 8 | 0 | 24
Participants
  Subjects with Any Complication | 8 | 7 | 7 |  | 22
  Acquired Sepsis | 2 | 2 | 2 |  | 5
  Apnea | 8 | 5 | 6 |  | 19
  Cystic Periventricular Leukomalcia | 0 | 0 | 0 |  | 1
  Patent Ductus Arteriosus | 3 | 3 | 4 |  | 10
  Pulmonary Hemorrhage | 1 | 0 | 1 |  | 1
  Intraventicular Hemorrhage | 0 | 1 | 3 |  | 4
  Necrotizing Enterocolitis | 1 | 1 | 1 |  | 1
  Retinopathy of Prematurity | 2 | 1 | 1 |  | 9

9. Other Pre Specified Outcome: nCPAP Failure Without Treatment Interruptions
Description: Number of subjects requiring mechanical ventilation or surfactant administration (nCPAP failure) but did not have a treatment interruption
Time Frame: Randomization to 72 Hours Post Randomization
Population: Intent-to-Treat Without Treatment Interruption
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg/kg | 75 mg/kg | 100 mg/kg | 150 mg/kg | nCPAP Alone
Number analyzed (Participants) | 7 | 3 | 6 | 0 | 24
Participants | 4 | 3 | 3 |  | 16

ADVERSE EVENTS:
Time Frame: From randomization to 36 weeks PMA
Description: This dose-escalation study was terminated after completion of the 100 mg/kg group for administrative purposes. No participants were enrolled in the 150 mg/kg group or received 150 mg/kg.
Arm/Group | 50 mg/kg | 75 mg/kg | 100 mg/kg | 150 mg/kg | nCPAP Alone
All-Cause Mortality (participants affected / at risk) | 1/8 | 1/8 | 0/8 | 0/0 | 0/24
Serious Adverse Events (participants affected / at risk) | 4/8 | 3/8 | 2/8 | 0/0 | 6/24
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 8/8 | 0/0 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50 mg/kg (N=8) | 75 mg/kg (N=8) | 100 mg/kg (N=8) | 150 mg/kg (N=0) | nCPAP Alone (N=24)
Anaemia neonatal (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 1 (1)
Sepsis neonatal (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 0
Hepatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1)
Laryngeal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) — Laryngeal trauma due to intubation
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) — Liver laceration
Intraventricular haemorrhage neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 (2) | 0 | 1 (1)
Necrotising enterocolitis neonatal (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 | 0 | 0 | 1 (1)
Neonatal respiratory distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 2 (2) | 0 | 0 | 1 (1)
Neonatal respiratory failure (Pregnancy, puerperium and perinatal conditions) | 0 | 1 (1) | 0 | 0 | 0
Apnoea neonatal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 (1)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 1 (1) | 0 | 2 (2)
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 1 (1) — Refractory shock
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50 mg/kg (N=8) | 75 mg/kg (N=8) | 100 mg/kg (N=8) | 150 mg/kg (N=0) | nCPAP Alone (N=24)
Anaemia neonatal (Blood and lymphatic system disorders) | 6 (6) | 4 (6) | 2 (2) | 0 (0) | 12 (16)
Bandaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 3 (3) | 3 (3) | 4 (4) | 0 (0) | 10 (10)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (13) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric hypomotility (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Salivary hypersection (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endotracheal intubation complication (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Inadvertent extubation
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oedema (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Methicillin-sensitive S. aureus (MSSA) colonization
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nosocomial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis neonatal (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blister (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Peripheral IV infiltration
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tracheal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anticonvulsant drug level above therapeutic level (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Increased levels of phenobarbital
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Coagulation time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 2 (3) | 4 (6) | 6 (11) | 0 (0) | 9 (11)
PO2 increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Reticulocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeding intolerance (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 4 (5)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypochloraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteopenia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periventricular leukomalacia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Agitation neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 5 (7) | 3 (5) | 0 (0) | 9 (9)
Fixed bowel loop (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraventricular haemorrhage neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 3 (3) | 1 (1) | 0 (0) | 11 (12)
Necrotising enterocolitis neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Neonatal respiratory distress syndrome (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 9 (12)
Periventricular haemorrhage neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinopathy of prematurity (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 9 (9)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Apnoea neonatal (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (5) | 6 (9) | 0 (0) | 19 (21)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasal mucosal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary interstitial emphysema syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Pulmonary oedema neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haemangioma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 4 (7)

LIMITATIONS AND CAVEATS:
The study was terminated prior to subject enrollment for the 150 mg TPL/kg dose by the sponsor for administrative reasons.

The overall results may have been impacted by treatment interruptions caused by clogging of study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The preparation and submittal for publication of a manuscript containing the study results shall be in accordance with a process determined by a mutual written agreement among Windtree Therapeutics, Inc. and participating institutions. The publication or presentation of any study results shall comply with all applicable privacy laws, including, but not limited to, HIPAA.

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-05-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT02528318/SAP_000.pdf
  • Study Protocol (2015-09-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT02528318/Prot_001.pdf